CLINICAL TRIAL: NCT07187726
Title: Multicenter Randomized Pivotal Stage Clinical Investigation Assessing the Communication of an Individualized AI-based Risk Prediction of Arm Lymphedema to Breast Cancer Patients With an Indication for Regional Lymph Node Irradiation and Their Physician as Part of Treatment Shared-decision
Brief Title: Arm Swelling Occurence in Breast Cancer Patients With Nodal Radiotherapy: Impact of Informing Them of AI-predicted Risk
Acronym: PRE-ACT-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UC-RAD-2407
Record Dates: First submitted 2025-06-21; First posted 2025-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Unilateral Breast Neoplasms
Keywords: Arm lymphedema; Individualized AI-based risk prediction
MeSH Terms: conditions — Unilateral Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication of the AI-based risk prediction to patient and physician. (Experimental)
  Interventions: Device: XAINET AI tool
- No communication of the AI-based risk prediction to patient and physician. (No Intervention)

INTERVENTIONS:
Device: XAINET AI tool — The AI-based prediction of arm lymphedema risk is communicated to the patient and treating physician.
  Arms: Communication of the AI-based risk prediction to patient and physician.

SUMMARY:
Radiotherapy after breast cancer surgery can lead to side effects like arm lymphedema (arm swelling). Lymphedema can cause long-term discomfort and affect quality of life.

The goal of this clinical investigation is to determine whether using an artificial intelligence (AI) tool to predict the risk of developing arm lymphedema after breast cancer radiotherapy can help patients and physicians make better treatment decisions.

This AI tool has been developed to determine each patient's personalized risk of developing lymphedema. The risk is shown using a web app that explains the factors involved and offers suggestions like using a compression sleeve to reduce the risk.

Women (≥18 years) with breast cancer (cT1-4, cN0-N3, M0) requiring regional lymph node irradiation post-mastectomy or breast-conserving surgery are eligible, regardless of hormone receptor status, tumor grade, or HER2 status.

Patients will be randomly divided into two groups:

* Experimental group: Patients and physicians will see the AI-predicted risk and use it to guide treatment choices.
* Control group: The risk is not shown.

The radiotherapy treatment will be exactly the same as the treatment that you would have received if you had not taken part in this clinical investigation. The only intervention will be whether or not the risk you are informed of the risk of developing lymphedema.

All patients will be followed for two years to monitor:

* How risk communication influences radiotherapy treatment choices
* The occurrence of side effects
* The predictive performance of the AI tool
* Patients' quality of life
* Compliance with compression sleeve use
* Loco-regional recurrence-free survival, distant disease-free survival, and overall survival

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent form prior to inclusion visit and to any study specific procedures
2. Women ≥ 18 years
3. Patients with unilateral invasive breast cancer, cT1-4, cN0-N3, M0 who had undergone radical surgery defined as mastectomy or breast conservation surgery with negative margins +/- (neo)-adjuvant systemic treatment. The patient can be included no matter the status of estrogen and progesterone receptors, malignancy grade, and HER2 status
4. Axillary lymph node staging (by axillary dissection or sentinel lymph node biopsy and/or marked lymph node biopsy [Marking Axillary lymph nodes with Radioactive Iodine seeds (MARI) procedure/ (Targeted Axillary Dissection (TAD) procedure] in case of neo-adjuvant systemic treatment) defining the indication for regional nodal irradiation to levels I+/- II+/- III+/- IV+/- interpectoral nodes (Rotter) +/- the IMC(Internal Mammary Chain)
5. ECOG performance status 0-2
6. Patient must be randomized within the recommended time period from last surgery or the last series of chemotherapy whichever comes last as per national or institutional guidelines in order not to delay radiotherapy treatment start
7. Women of childbearing potential must agree to use adequate contraception for the duration of study participation and up to 3 months following completion of radiotherapy
8. Patient is willing and able to comply with the protocol for the duration of the clinical investigation including undergoing treatment and scheduled visits, and examinations including follow-up
9. Patient affiliated to or a beneficiary of the local social security system, health service or other local regulatory requirements

Exclusion Criteria:

1. Previous breast cancer or Ductal Carcinoma in Situ (DCIS) of the ipsilateral breast
2. Bilateral breast cancer
3. Patient with previous non-breast malignancy, with the exception of cancer in complete remission for over 5 years and low risk of recurrence. Patients with the following diseases can be accepted despite less than 5 years disease free interval: carcinoma in situ of the cervix, melanoma in situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin
4. Patient who has an indication for boost to one or more regional nodes
5. Previous radiation therapy to the chest region
6. Patients having arm swelling requiring arm sleeve prescription at baseline
7. Any condition that prevents the patient from wearing a compression sleeve for 8h/day from the first day of radiation therapy until 3 months after the initiation of adjuvant radiotherapy
8. Pregnant or breastfeeding women
9. Patient already included in another therapeutic study involving radiotherapy dose/regimen/technique and/or arm lymphedema risk
10. Person deprived of their liberty or under protective custody or guardianship
11. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Arm lymphedema | At 2 years
  Cumulative incidence of arm lymphedema on the treated side 2 years after adjuvant radiotherapy. The definition of arm lymphedema is ≥5% increased arm circumference measured 15 cm proximal and/or 10 cm distal of the olecranon of the treated side from baseline, compared to the contralateral side circumference and to its baseline value

SECONDARY OUTCOMES:
Impact of communicating the risk prediction for arm lymphedema on the choice of radiotherapy modality, fractionation, technique and nodal levels irradiated | Up to 3 months from randomization.
  Radiotherapy modalities: technique used, fractionation (use of moderately and ultra-hypofractionated), and lymph node levels treated will be compared in both arms
Acute and late toxicity during the study | Throughout study completion, up to 2 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders
Range of shoulder motion (ROM) of the arms | Throughout study completion, up to 2 years.
  The range of shoulder motion (ROM) of the arms (flexion/abduction) will be reported by the radiation oncologist according to a circular scale
Breast cosmetic result | Throughout study completion, up to 2 years.
  The global cosmetic result after breast conservation surgery will be based on Harris 4-point scale (4-point Likert scale: Excellent, Good, Fair, Poor)
Performance of the arm lymphedema risk prediction model | At 2 years
  The performance will be assessed by the discrimination and the calibration of the model in the control arm. The discrimination refers to how well the model differentiates patients at higher risk of having an event from those at lower risk. For assessing discrimination at fixed time point of occurrence of event of interest, the area under the receiver operating characteristic curve (AUC) will be calculated. The calibration expresses the agreement between the observed and predicted outcome values. To assess whether the observed event rate equals the predicted risk in different groups of predicted risks, calibration curve will be created.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, end of treatment visit, 1 year and 2 years
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level
Quality of Life Questionnaire - Breast cancer module (QLQ-BR23) | At baseline, end of treatment visit, 1 year and 2 years
  This EORTC breast cancer specific questionnaire is intended to supplement the QLQ-C30.
  The QLQ-BR23 contains 23 items incorporating five multi-item scales to assess systemic therapy side effects, arm symptoms, breast symptoms, body image and sexual functioning. In addition, single items assess sexual enjoyment, hair loss and future perspective. All items are rated on a four-point Likert-type scale (1 = "not at all", 2 = "a little", 3 = "quite a bit", and 4 = "very much"), and are linearly transformed to a 0-100 scale. For all items but sexual functioning and sexual enjoyment, higher scores indicate more severe symptoms
The Developed 5-level version of EQ-5D (EQ-5D-5L) questionnaire | At baseline, end of treatment visit, 1 year and 2 years
  Developed by the EuroQol group, the self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials consists of a descriptive system and a visual analogue scale (VAS) The EQ-5D-5L descriptive system comprises five dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each dimension has 5 levels (1 = "no problems", 2 = "slight problems", 3 = "moderate problems", 4 = "severe problems", and 5 = "extreme problems"). This questionnaire provide a 5-digit score which generate a health state profile. The VAS records the patient's self-rated health on a vertical visual analogue scale where the score range from 0 (The best health you can image) to 100 (The worst health you can image). The VAS is used as a quantitative measure of health outcome that reflects the patient's own judgement
Compliance with compression arm sleeve use | At end of treatment visit, 3-month after starting radiotherapy, at 1 year and 2 years
  Compliance with the use of the compression arm sleeve will be measured by the frequency with which the patient wears it according to the patient
Loco-regional relapse-free survival (RFS) | From randomization until the first invasive ipsilateral breast tumor recurrence, loco regional invasive recurrence, ipsilateral DCIS or death from any cause up to 2 years
  Locoregional recurrence-free survival is the time from randomisation until locoregional recurrence (as the first recurrence event) or death
Distant disease-free survival (DDFS) | From randomization until the recurrence of disease or death from any cause up to 2 years
  Distant disease-free survival is defined as the time from randomization until the recurrence of disease (first, occurrence of metastasis or distant relapse) or death from any cause using DATECAN definitions of breast-cancer related endpoints
Overall survival (OS) | From randomization to death from any cause, up to 2 years
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Centre Marie Curie, Arras
  - Centre Pierre Curie, Beuvry
  - Clinique Tivoli Ducos, Bordeaux
  - ROC 37, Chambray-lès-Tours
  - CHI Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Guillaume Le Conquérant, Le Havre
  - Centre Antoine Lacassagne, Nice
  - Institut Godinot, Reims
  - ICO Nantes Saint Herblain, Saint-Herblain
  - Institut de Cancérologie Strasbourg Europe, Strasbourg
  - Gustave Roussy, Villejuif